CLINICAL TRIAL: NCT02235571
Title: iChoose Kidney Decision Aid for Treatment Options Among End-Stage Renal Disease (ESRD) Patients
Brief Title: iChoose Decision Kidney Aid for End-Stage Renal Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Columbia University (Other); Northwestern University (Other); Satellite Healthcare (Other); Norman S. Coplon Extramural Grant Program (Unknown)
Responsible Party: Principal Investigator, Rachel Patzer, PhD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00076067
Record Dates: First submitted 2014-09-06; First posted 2014-09-10 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: End-Stage Kidney Disease; Kidney Failure, Chronic; Kidney Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): These subjects are receiving standard patient education
- iChoose Kidney Decision Aid (Experimental): These subjects receive iChoose Kidney Decision Aid along with standard patient education
  Interventions: Behavioral: iChoose Kidney Decision Aid

INTERVENTIONS:
Behavioral: iChoose Kidney Decision Aid — Providers will use a shared decision making tool with patients via iPhone, iPad, or web which explains predicted individualized risk of mortality on dialysis vs. transplant during the evaluation appointment for kidney transplant.
  Arms: iChoose Kidney Decision Aid

SUMMARY:
The investigators developed iChoose Kidney -- a shared decision-making support tool accessible through iPad, iPhone, or the web -- to provide ESRD patients and their providers with a simple, standardized, easily accessible, statistically robust tool for use in the clinic to guide patient education and healthcare decision-making about treatment options of dialysis or kidney transplantation. The iChoose Kidney decision aid provides patients with estimates of their individualized 1 and 3-year risks of mortality on dialysis vs. transplantation, based on previous national data. The tool has the potential to improve communication and decision-making between patients and their healthcare providers and improve access to kidney transplantation among patients with ESRD.

This will be a two-arm, randomized study, and will be conducted at 3 large transplant centers with diverse patient populations. One group of patients will receive standard education alone during their scheduled transplant evaluation. The second group will receive the standard education as well have the provider use the iChoose Kidney aid with them. The project timeline will be a total of 24 months inclusive of enrollment, follow-up, data analysis, and outcome evaluation.

This study will assess how well the iChoose decision aid works in improving patient knowledge, preferences for treatment, and patient access to transplant. The study will also assess whether providers find the tool useful for providing ways to share information with patients about ways to treat their kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of end-stage renal disease (ESRD) and on dialysis for < 1 year
* English-speaking
* Subjects coming in for transplant medical evaluation
* Age > 18 years

Exclusion Criteria:

* Severe cognitive or visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2014-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the iChoose Kidney intervention to improve knowledge and shared decision-making between patients and physicians regarding ESRD treatment options. | Up to 19 months
  Patient knowledge of the survival benefit of transplant and the patient's individualized mortality risk

SECONDARY OUTCOMES:
Patient access to transplant | Up to 19 months
  Evaluation completion, waitlisting, transplant

OTHER OUTCOMES:
Patient treatment preferences | Up to 19 months
  Patient preference for transplant vs. dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Patzer, PhD, MPH, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Transplant Center, Atlanta, Georgia
  - Northwestern University (Kovler Transplant Center), Chicago, Illinois
  - Columbia University Medical Center, New York, New York

REFERENCES:
- [Derived] Patzer RE, McPherson L, Basu M, Mohan S, Wolf M, Chiles M, Russell A, Gander JC, Friedewald JJ, Ladner D, Larsen CP, Pearson T, Pastan S. Effect of the iChoose Kidney decision aid in improving knowledge about treatment options among transplant candidates: A randomized controlled trial. Am J Transplant. 2018 Aug;18(8):1954-1965. doi: 10.1111/ajt.14693. Epub 2018 Mar 26. PMID 29446209